CLINICAL TRIAL: NCT04707352
Title: Impact on Atrial Remodeling of Dapaglifozin in Patients With Heart Failure .
Acronym: MODA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-20594 - MODA study
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Interventional, open-label and single-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dapagliflozin (Experimental): The baseline procedures will be performed on the same day of screening or within the next five working days. All the baseline procedures will be performed on the same day. The baseline procedures include biobank, clinical assessment and echocardiogram, on the same day. In the following 24 hours, the patient will initiate Dapagliflozin at the recommended dose of 10 mg daily during 6 months. Temporary discontinuation may be considered at investigator criteria as in cases of symptomatic hypotension or acute declines in renal function and after discarding other potential causes.
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — All eligible subjects will receive Dapagliflozin 10 mg each day. The study treatment will be provided for the duration of the trial from baseline (Day 1) through last visit (Day 180).

SUMMARY:
Dapagliflozin reduces the risk of de novo heart failure (HF) in diabetics and, recently, it has shown to improve the prognosis of patients with HF and reduced left ventricular ejection fraction (HFrEF), by preventing HF decompensations and cardiovascular death. The benefit showed by dapagliflozin in HFrEF was irrespective of diabetes status and glycemic control, which raises the question of which mechanisms are underlying apart from SGLT2 inhibition. In addition, the impact of dapagliflozin on cardiac remodeling parameters, as assessed by echocardiography and biomarkers, is not well established. In particular, left atrial (LA) remodeling represents a relevant prognostic marker, which has received a greater attention in the last years in the context of new imaging tools.

The purpose of this study is to assess the effect of dapagliflozin therapy over a period of 6 months in LA remodeling parameters, including geometry and function, as well as complementary biomarkers in patients with chronic HF regardless left ventricular ejection fraction (LVEF). This protocol will allow for evaluation of improved understanding of the interplay between dapagliflozin and LA function , biomarkers, remodeling and outcomes, and will carefully assess such relationships within important cohorts of subjects, such as those with reduced and preserved LVEF.

This protocol will also generate a biorepository of well-handled and carefully considered biomarkers, which will allow a better understanding of dapagliflozin mechanism of action.

DETAILED DESCRIPTION:
The reduction of death and HF related events observed with dapagliflozin make necessary to clarify the mechanisms underlying these clinical benefits. Currently, dapagliflozin is indicated in patients with diabetes irrespective of the presence of HF. The initiation in patients with HF represents an opportunity to elucidate the effect of dapagliflozin on cardiac remodeling in this population. Therefore, we propose a study that aims to assess the effects of dapagliflozin in echocardiographic parameters of cardiac remodeling, with special interest in LA geometry and function, as well as in biomarkers reflecting expanded pathophysiological pathways. LA volume has shown to identify the progression of HF irrespective of LVEF and, therefore, it represents a meaningful measure of the cardiac impact of dapagliflozin in the entire spectrum of chronic HF.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

  * Prior diagnosis of HF, with at least one hospitalization for HF at any time.
* NYHA class I-IV.
* LVEF available (echocardiogram or cardiac MRI) within the last 12 months prior to enrolment.
* Treatment according with contemporary guidelines recommendations and with stable doses of oral loop diuretics for at least 4 weeks
* NT-proBNP >600 pg/ml at screening (≥400 pg/ml if hospitalized for HF within the previous 12 months; ≥900 pg/ml If concomitant AF at
* Screening irrespective of time to last HF hospitalization).

Exclusion Criteria:

* Dapagliflozin or other SGLT2i at any time in prior 6 months.
* Type 1 diabetes mellitus (T1D)
* Estimated glomerular filtration rate < 30 ml/min/1.73 m2 as measured by the simplified Modification of Diet in Renal Disease (MDRD) formula at screening.
* Symptomatic hypotension or systolic blood pressure (SBP) <95 mmHg on 2 consecutive measurements at screening.
* Uncontrolled hypertension, defined as SBP >160 mmHg.
* Current acute decompensated HF or hospitalization due to decompensated HF within 4 weeks prior to enrolment
* The use of outpatient or inpatient i.v. diuretic therapy within 4 weeks prior to baseline.
* Subjects who are currently receiving or have received inotropic agents within 12 weeks prior to baseline.
* Myocardial infarction, unstable angina, stroke or transient ischemic attack within 12 weeks prior to enrolment
* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting or valvular repair/replacement within 12 weeks prior to enrolment or planned to undergo any of these operations after inclusion
* Implantation of a cardiac resynchronization therapy (CRT) within 12 weeks prior to enrolment or intent to implant a CRT device
* Previous cardiac transplantation or implantation of a ventricular assistance device (VAD) or similar device, or implantation expected after inclusion
* HF due to restrictive cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy or uncorrected primary valvular disease
* Symptomatic bradycardia or second or third degree heart block without a pacemaker
* History of allergic reactions or intolerance to dapagliflozin, or other iSGLT2, or any other compound
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within one year.
* Hepatic impairment aspartate transaminase [AST] or alanine transaminase [ALT] >3x the upper limit of normal [ULN]; or total bilirubin >2x ULN at time of screening)
* Women of child-bearing potential (ie, those who are not chemically or surgically sterilised or who are not post-menopausal) who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator or women who have a positive pregnancy test at enrollment or randomization or women who are breast-feeding
* Participation in another clinical trial during the last month prior to enrolment
* Inability of the patient, in the opinion of the investigator, to understand and/or comply with study medications, procedures and/or follow-up or any conditions that, in the opinion of the investigator, may render the patient unable to complete the study
* Any concomitant disease limiting life expectancy in the following year (other than heart failure)
* No possibility to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-03-26 (Actual); Study Completion 2023-03-26 (Actual)

PRIMARY OUTCOMES:
Change in LAVI from baseline to 6 months. | Up to 6 months

SECONDARY OUTCOMES:
Change in LAVI-min (minimal left atrial volume index) | Up to 6 months
Change in LAEF (left atrial ejection) | Up to 6 months
Change in LAFI (left atrial functional index) | Up to 6 months
Change in LA reservoir, conduit and pump volumes, emptying fractions and strain rates | Up to 6 months
Change in Left ventricular end-systolic volume index (LVESVi) | Up to 6 months
Change in left ventricular mass index (LVMI) Change in ventricular end-diastolic volume index (LVEDVi) | Up to 6 months
Change in global longitudinal strain (GLS) | Up to 6 months
Change in tricuspid annular plane systolic | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Domingo Pascual Figal, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Hospital Clinico Universitario Virgen de la Arrixaca, Murcia, Spain

REFERENCES:
- [Derived] Pascual-Figal DA, Zamorano JL, Domingo M, Morillas H, Nunez J, Cobo Marcos M, Riquelme-Perez A, Teis A, Santas E, Caro-Martinez C, Pinilla JM, Rodriguez-Palomares JF, Dobarro D, Restrepo-Cordoba MA, Gonzalez-Juanatey JR, Bayes Genis A; DAPA-MODA Study Investigators. Impact of dapagliflozin on cardiac remodelling in patients with chronic heart failure: The DAPA-MODA study. Eur J Heart Fail. 2023 Aug;25(8):1352-1360. doi: 10.1002/ejhf.2884. Epub 2023 Jun 7. PMID 37211950